CLINICAL TRIAL: NCT00030459
Title: Randomized Feasibility Study Of Active Symptom Control With Or Without Chemotherapy In The Treatment Of Patients With Mesothelioma
Brief Title: Palliative Therapy With or Without Chemotherapy in Treating Patients With Malignant Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Thoracic Society (Other)
Collaborators: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: BTS-MESO-1; CDR0000069167 (Registry Identifier: PDQ (Physician Data Query)); MRC-BTS-MESO-1; EU-20134
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2003-05

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; Mitomycin; Vinblastine; Vinorelbine

INTERVENTIONS:
Drug: cisplatin
Drug: mitomycin C
Drug: vinblastine sulfate
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Palliative therapy may help patients with advanced cancer live more comfortably. It is not yet known if palliative therapy is more effective with or without chemotherapy in treating patients who have malignant mesothelioma.

PURPOSE: Randomized phase II trial to compare the effectiveness of palliative therapy with or without different chemotherapy regimens in treating patients who have malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of palliative therapy alone versus palliative therapy with mitomycin, vinblastine, and cisplatin versus palliative therapy with vinorelbine in patients with malignant mesothelioma.
* Determine the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of three treatment arms.

* Arm I: Patients receive palliative therapy alone comprising non-chemotherapeutic therapy (e.g., radiotherapy, painkillers, steroids, relaxants, and special pain relief techniques).
* Arm II: Patients receive palliative therapy as in arm I and chemotherapy comprising mitomycin IV (courses 1, 2, and 4 only), vinblastine IV, and cisplatin IV over 4 hours on day 1. Chemotherapy repeats every 21 days for a total of 4 courses.
* Arm III: Patients receive palliative therapy as in arm I and chemotherapy comprising vinorelbine IV over 5 minutes once weekly on weeks 1-6 and 9-14.

Quality of life is assessed at baseline for all patients; at weeks 3, 6, 9, and 12 for arm I; at weeks 4, 7, 10, and 13 for arm II; at weeks 3, 6, 10, and 13 for arm III; at weeks 21 and 29, and then every 8 weeks thereafter for all patients.

Patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 60 patients (20 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Immunohistochemically or cytologically confirmed malignant mesothelioma

  * Epithelial and other histological types
* Symptomatic pleural effusion allowed if treated and controlled by drainage, pleurodesis, or pleurectomy
* Prior surgical resection allowed if stable or progressive disease by 2 CT scan measurements at least 6 weeks apart

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm3
* Neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Considered medically fit to receive chemotherapy
* No other disease or prior malignancy that would preclude study
* No clinical evidence of infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for mesothelioma

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Overall Officials: Martin F. Muers, MD, Study Chair — Leeds General Infirmary; David J. Girling, MD, Study Chair — Medical Research Council
Locations (9):
- United Kingdom (9):
  - Princess Royal Hospital, Hull, England
  - Leeds Teaching Hospital Trust, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Medical Research Council Clinical Trials Unit, London, England
  - Royal Marsden Hospital, Sutton, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Stobhill General Hospital, Glasgow, Scotland
  - Dorothy House Foundation, Bradford-Onavon
  - St. Peters Hospital, Chertsey Surrey